CLINICAL TRIAL: NCT00768963
Title: Ranibizumab for the Inhibition of Neovascularization in Pterygia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Sonia Yoo, Professor, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20080012
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Pterygium
Keywords: ranibizumab; pterygium
MeSH Terms: conditions — Pterygium | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients will receive one injection of ranibizumab 3 days prior to surgery
  Interventions: Drug: ranibizumab
- 2 (Experimental): Patients will undergo one injection of ranibizumab at the time of surgery
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab — 0.5 mg subconjunctival ranibizumab 3 days prior to surgery
  Other Names: Lucentis
  Arms: 1
Drug: ranibizumab — 0.5 mg subconjunctival ranibizumab at the time of surgery
  Other Names: Lucentis
  Arms: 2

SUMMARY:
The primary purpose of this trial is to evaluate the safety and tolerability of ranibizumab given via subconjunctival injection in patients undergoing pterygium surgery.

DETAILED DESCRIPTION:
As a secondary objective, this study also aims to establish the tissue concentration of ranibizumab when delivered via subconjunctival injection in patients undergoing pterygium excision and to determine the effects of ranibizumab on conjunctival healing, corneal epithelial healing, and wound dehiscence.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible if the following criteria are met:
* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 18 years
* Patient related considerations: All patients of both genders will be considered for enrollment.
* Disease related considerations:

  * Patients with pterygia will be considered for enrollment if the pterygium meets standard pterygium excision criteria including encroachment into the visual axis
  * severe induced astigmatism
  * foreign body sensation unresponsive to medical therapy.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from this study:

* Pregnancy (positive pregnancy test)
* Women seeking to become pregnant
* Lactating women
* Prior enrollment in the study
* Prior glaucoma surgery in the region of the pterygium
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-10; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The primary purpose of this trial is to evaluate the safety and tolerability of ranibizumab given via subconjunctival injection in patients undergoing pterygium surgery. | 2 years

SECONDARY OUTCOMES:
This study aims to establish the tissue concentration of ranibizumab when delivered via subconjunctival injection and determine the effects of ranibizumab on conjunctival healing, corneal epithelial healing, and wound dehiscence. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Yoo, MD, Principal Investigator — Bascom Palmer Eye Institute
Locations (1):
- Bascom Palmer Eye Institute, Miami, Florida, United States

REFERENCES:
- [Derived] Galor A, Yoo SH, Piccoli FV, Schmitt AJ, Chang V, Perez VL. Phase I study of subconjunctival ranibizumab in patients with primary pterygium undergoing pterygium surgery. Am J Ophthalmol. 2010 Jun;149(6):926-931.e2. doi: 10.1016/j.ajo.2010.01.015. Epub 2010 Apr 24. PMID 20417925